CLINICAL TRIAL: NCT03516773
Title: An Evaluation of the Pharmacokinetics and Pharmacodynamics of Oral Parathyroid Hormone [PTH (1-34)] and NATPARA® in Patients With Hypoparathyroidism
Brief Title: Oral PTH(1-34) PK and PD Study in Patients With Hypoparathyroidism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Entera Bio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ENT-04-2018
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Hypoparathyroidism
Keywords: Hypoparathyroidism, PTH(1-34), Parathyroid Hormone
MeSH Terms: conditions — Hypoparathyroidism | interventions — Parathyroid Hormone

STUDY DESIGN:
Intervention Model Description: Randomized, active comparator, two-part, within-part, partial crossover design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment A (Experimental): Intervention: EB612 (EBP05) 2.25 mg orally (PO) four times a day (QID) (approximately 5 hours apart) for 4 doses, for a total dose of 9 mg per day
  Interventions: Drug: EB612 (EBP05)
- Treatment B (Experimental): Intervention: EB612 (EBP05) 2.25 mg PO twice a day (BID) (approximately 10 hours apart) for 2 doses, for a total dose of 4.5 mg per day
  Interventions: Drug: EB612 (EBP05)
- Treatment C (Active Comparator): Intervention: NATPARA/NATPAR PTH(1-84) 100 μg subcutaneous injection once daily (single dose)
  Interventions: Drug: NATPARA/NATPAR
- Treatment D (Experimental): Intervention: EB612 (EBP05) 2.25 mg PO TID (dose 1 and dose 2 approximately 10 hours apart; dose 2 and dose 3 approximately 5 hours apart- TID schedule option 2), for a total dose of 6.75 mg per day
  Interventions: Drug: EB612 (EBP05)
- Treatment E - EB612 (EBP05) (Experimental): Intervention: EB612 (EBP05) 0.75 mg PO TID (dose 1 and dose 2 approximately 10 hours apart; dose 2 and dose 3 approximately 5 hours apart- TID schedule option 2), for a total dose of 2.25 mg per day
  Interventions: Drug: EB612 (EBP05)

INTERVENTIONS:
Drug: EB612 (EBP05) — Entera Bio's proprietary drug for the administration of PTH(1-34) orally
  Other Names: Oral PTH(1-34)
  Arms: Treatment A; Treatment B; Treatment D; Treatment E - EB612 (EBP05)
Drug: NATPARA/NATPAR — A PTH replacement (PTH [1-84]; NATPARA (Shire-NPS Pharmaceuticals, Inc., Lexington, Massachusetts) was approved by the United States (US) Food and Drug Administration (FDA) in April 2015 / NATPAR (Shire Pharmaceuticals Ltd., Dublin, Ireland) was approved by the European Medicines Agency in April 2017 for use as an adjunct to calcium and vitamin D to control hypocalcemia in patients with hypoparathyroidism. Like many other hormonally active peptides, PTH (1 84); NATPARA is parenterally administered. In this protocol when a specific formulation is referenced (e.g. NATPARA) it may be read interchanged with the alternate formulation (e.g. NATPAR).
  Other Names: PTH(1-84)
  Arms: Treatment C

SUMMARY:
A Randomized, active comparator, two-part, partial crossover design. The study is designed to assess the pharmacokinetics and pharmacodynamics of EnteraBio's Oral PTH(1-34) [EB612 (EBP05)] in adult patients with hypoparathyroidism.

ELIGIBILITY:
-Criteria for Inclusion:

1. Confirmed diagnosis of primary hypoparathyroidism, as defined by the European Society of Endocrinology as a patient with hypocalcemia and inappropriately low PTH levels. If the source of hypoparathyroidism is surgical or iatrogenic, diagnosis must be for more than 1 year. If the source of hypoparathyroidism is not surgical or iatrogenic, and confirmed by inappropriately low PTH levels and hypercalciuria, diagnosis does not have time limitations.
2. 1, 25(OH)2D levels ≥20 ng/mL.
3. Signed Informed Consent Form).
4. Age 18 to 80 years with body mass index of 19 to 35 kg/m2.
5. Patients able to adhere to the visit schedule and protocol requirements.

Criteria for Exclusion:

1. Known history of hypoparathyroidism resulting from an activating mutation in the calcium sensing receptor gene or impaired responsiveness to PTH (pseudohypoparathyroidism).
2. Hemoglobin <11.5 g/dL (females) / <12.5g/dL (males) [lower limit of reference range, 12 to 15 g/dL and 13 to 17 g/dL]
3. Acute or chronic renal failure (estimated glomerular filtration rate <60 mL/min/1.73 m²).
4. Significant liver function impairment (liver enzymes above ×2 the upper limit of normal range).
5. Patients with hypomagnesemia should be excluded unless serum magnesium is corrected prior to study initiation.
6. Active gastrointestinal inflammatory, gastrointestinal motility disorders, and chronic gastritis, such as ulcerative colitis, Crohn's disease, irritable bowel syndrome, short bowel syndrome, celiac disease, gastroparesis, etc.
7. Active hepatitis or acquired immunodeficiency syndrome (AIDS)/AIDS-related syndrome
8. Any conditions or factors that, in the judgment of the Investigator, somehow may impact gastrointestinal absorption.
9. Concurrent therapy with the following medications: (1) 14 days: thiazide diuretics; loop diuretics (2) 30 days: lithium, systemic corticosteroid; (3) 1 month: calcitonin, cinacalcet hydrochloride, recombinant PTH(1-84) or N-terminal PTH or PTH-related peptide fragments or analogs; (4) females only; changes in hormone replacement therapy within 2 months; (5) 3 months: methotrexate, growth hormone, digoxin; raloxifene or similar selective estrogen receptor modulators; (7) chronic or concurrent use of gastrointestinal motility modulators (domperidone, loperamide, erythromycin metoclopramide etc.); and (8) other concurrent therapy that, in the Investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study medication.
10. Significant drug or alcohol abuse as assessed by the PI.
11. Treatment with any investigational product within the last 30 days or 5 half-lives (if known) whichever is longer.
12. Has participated as a patient in any investigational drug study within the last 30 days preceding the screening visit or plans to participate in another investigational drug study at any time during the study or within 30 days of his/her completion of this study.
13. Presence of any other condition or circumstance that, in the judgment of the Investigator, might increase the risk to the patient or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.
14. Historical documented allergy to soy bean products or known hypersensitivity to the PTH (1-34).
15. Patients at increased risk for osteosarcoma, such as those with Paget's disease of bone or unexplained elevations of alkaline phosphatase, hereditary disorders predisposing to osteosarcoma, or with a prior history of external beam or implant radiation involving the skeleton.
16. Patients with skeletal malignancies or bone metastases.
17. Pregnancy or suspected pregnancy or lactating. Female patients of childbearing potential must have a negative pregnancy test at screening and be willing and able to use two medically acceptable methods of birth control (reliable use of oral contraceptive with physical barrier, non-hormonal intrauterine device with condom, diaphragm with condom, or condom with spermicide) from the screening visit through 90 days from last dose or declare that they are abstaining from sexual intercourse from the screening visit through the study termination visit or are surgically sterile (have undergone bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) or postmenopausal. True abstinence can only be in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, and postovulation methods), declaration of abstinence for the duration of a study, and withdrawal are not acceptable methods of contraception.

Childbearing potential is defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal. Women will be defined as postmenopausal if they have been amenorrheic for 12 months (prior to signature of Informed Consent Form) without an alternative medical cause.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-17 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2019-02-24 (Actual)

PRIMARY OUTCOMES:
Plasma PTH(1-34) levels | 18 weeks
  Pharmacokinetic Parameter
Serum albumin-adjusted total calcium levels | 18 weeks
  Pharmacodynamic Parameter
urinary calcium levels | 18 weeks
  Pharmacodynamic Parameter

SECONDARY OUTCOMES:
Adverse Events | 60 days
  Safety Parameter
Rate of Adverse Events leading to discontinuation | 60 days
  Tolerability Parameter

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Santora, MD, Study Chair — Entera Bio Ltd.
Locations (1):
- Clinical Research Center Hadassah Ein Kerem Medical Center, Jerusalem, Israel